CLINICAL TRIAL: NCT05855668
Title: Phenotyping Patients With Alcohol and Cannabis Use Disorders Using the Addictions Neuroclinical Assessment
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); AFP Innovation Fund (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021/085
Record Dates: First submitted 2023-05-04; First posted 2023-05-11 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Alcohol Use Disorder; Cannabis Use Disorder
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Alcohol Use Disorder (Other): Participants will be treated with 12 weeks of CBT for AUD (group therapy) and have the option to receive evidence-based pharmacotherapy for AUD guided by a pharmacotherapy algorithm.
  Interventions: Behavioral: CBT
- Cannabis Use Disorder (Other): Participants will be treated with 12 weeks of CBT + motivational enhancement therapy for CUD (group therapy).
  Interventions: Behavioral: CBT

INTERVENTIONS:
Behavioral: CBT — 12 weeks of group CBT for AUD or CUD

SUMMARY:
This 2-arm study will recruit participants with 1) alcohol use disorder and 2) cannabis use disorder for a 12-week cognitive behavioral therapy, following a thorough baseline assessments on executive function, incentive salience, and negative emotionality.

DETAILED DESCRIPTION:
Although effective evidence-based interventions have been developed for alcohol and cannabis use disorders, it is still unclear which individuals respond best to treatment. A recent model known as the Addictions Neuroclinical Assessment (ANA) proposes that assessing for differences in three neurofunctional domains (executive function, incentive salience, and negative emotionality) could allow for a stronger neuroscience-based framework for understanding heterogeneity in response to addiction treatments but this has never been tested prospectively. In this study, we will recruit two groups: (1) participants with alcohol use disorder (AUD) and (2) participants with cannabis use disorder (CUD). Participants will undergo thorough baseline assessments of each of the three ANA domains prior to evidence-based treatment for their respective disorders. Individuals with AUD will be treated with 12 weeks of cognitive behavioral therapy (CBT) for AUD plus optional pharmacotherapy guided by a pharmacotherapy algorithm. Individuals with CUD will be treated with 12 weeks of CBT + motivational enhancement therapy for CUD. The primary objective of the study is to assess whether baseline ANA measures are associated with changes in drug consumption and craving over treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Patient has been referred to or intends to participate in either the AUD or CUD Integrated Care Pathway (and is therefore willing to participate in group psychotherapy).
2. Able to communicate and provide informed consent in English.
3. 18 years of age or older.
4. Willing and able to safely abstain from substances (other than nicotine or tobacco products), including alcohol and cannabis, for 12 hours prior to the eligibility and task-based assessments.
5. Meets DSM-5 diagnostic criteria for AUD (AUD group) or CUD (CUD group)
6. Meets criteria for risky drinking, defined as > 10 drinks per week for females and > 15 drinks per week for males on average over the past 30 days (AUD group) or daily or near-daily cannabis use over the past 30 days, defined as ≥ 4 days of cannabis use per week on average (CUD group)

Exclusion Criteria:

1. Active suicidal ideation at time of assessment.
2. Suicide attempt within the past month.
3. Unstable psychiatric or medical status (e.g., acute psychosis or mania) or unstable use of another substance that may interfere with participation in groups (e.g. active fentanyl use).
4. Enrollment in another study that conflicts with the procedures or scientific integrity of this study.
5. Individuals planning to be out of the province for a substantial amount of time during the treatment period will not be permitted to enroll.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2022-11-10 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Change in Number of Binge Drinking Days During Treatment Assessed by the Timeline Followback Interview (TLFB) (AUD Group) | 12 weeks
  Number of binge drinking days (≥ 4 drinks during a single day for females, ≥ 5 drinks during a single day for males)
Change in Cannabis Use Frequency During Treatment Assessed by the Timeline Followback Interview (TLFB) (CUD group) | 12 weeks
  Number of days per week in which individuals used cannabis
Change in Average Drinks Per Day During Treatment Assessed by the Timeline Followback Interview (TLFB) (AUD Group) | 12 weeks
  Average number of drinks per day
Change in Amount of Cannabis Used Per Week (grams/week) During Treatment Assessed by the Timeline Followback Interview (TLFB) (CUD group) | 12 weeks
  Amount of cannabis used per week
Change in Self-Reported Alcohol Craving During Treatment Assessed by the Penn Alcohol Craving Scale (PACS) (AUD Group) | 12 weeks
  Measures craving for alcohol (minimum score = 0; maximum score = 30; higher score indicates greater levels of craving)
Change in Self-Reported Cannabis Craving During Treatment Assessed by the Marijuana Craving Questionnaire-Short Form (MCQ) (CUD Group) | 12 weeks
  Measures craving for marijuana (minimum score = 17; maximum score = 119; higher score indicates greater levels of craving)

SECONDARY OUTCOMES:
Retention in Treatment (AUD and CUD groups) | 12 weeks
  Proportion of study participants that complete the treatment. Individuals who miss their first 2 sessions of therapy or miss more than 3 sessions of psychotherapy (i.e. ≥ 4 sessions or 33% of sessions) will be considered to have dropped out of treatment and will be discharged from the program. Participants who do not show up to any groups will not be included in this or other analyses.
Change in Depressive Symptoms during Treatment Assessed Using the Patient Health Questionnaire-9 (PHQ-9) (AUD and CUD groups) | 12 weeks
  Measures depressive symptoms (minimum score = 0; maximum score = 27; higher scores indicate higher levels of depressive symptoms)
Change in Anxiety Symptoms During Treatment Using the Generalized Anxiety Disorder-7 (GAD-7) (AUD and CUD groups) | 12 weeks
  Measures generalized anxiety (Minimum score = 0; maximum score = 21; higher scores indicate higher levels of anxiety)
Change in Quality of Life During Treatment Assessed Using the Abbreviated World Health Organization Quality of Life Scale (WHOQOL-BREF) (AUD and CUD Groups) | 12 weeks
  Measures quality of life (scores are transformed to 0-100; higher scores indicate higher quality of life)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Sloan, MD, Principal Investigator — Centre for Addiction and Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No